CLINICAL TRIAL: NCT04180306
Title: Implementation of Pediatric Early Warning Scores and a Context-adapted Resuscitation Training Course to Improve Outcomes in an LMIC Pediatric Inpatient Oncology Ward
Brief Title: PEWS Implementation in an LMIC Setting
Acronym: PEWSPAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Michelle Niescierenko, Attending Physician, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PEWSpalestine
Record Dates: First submitted 2019-11-23; First posted 2019-11-27 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inpatient pediatric oncology patients (Other): All patients admitted to the pediatric oncology ward will be in the cohort
  Interventions: Other: pediatric early warning scoring system and resuscitation curriculum

INTERVENTIONS:
Other: pediatric early warning scoring system and resuscitation curriculum — teaching resuscitation to medical providers and implementing a scoring tool to help identify patients at risk for clinical deterioration in an inpatient setting

SUMMARY:
The PEWS implementation study will be undertaken with the following objectives:

1. Assess the effectiveness of implementation of PEWS and resuscitation training to identify patients at risk for clinical deterioration and to impact the frequency of clinical interventions made by treating providers on these patients.
2. Assess the effectiveness of implementation of PEWS and resuscitation training to impact time sensitive clinical interventions made on patients at risk for clinical deterioration.
3. Assess the impact of implementation of PEWS and resuscitation training on length of stay for patients admitted to the pediatric oncology ward.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for the study are defined as pediatric patients (between birth and 12 years of age) admitted and subsequently discharged from the pediatric oncology ward in Beit Jala, Palestine and Gaza City, Palestine between March 2019 to June 2020

Exclusion Criteria:

* Patients will be excluded if they are not admitted to inpatient status. No oncology outpatients such as those in the infusion program will be included.

Ages: 0 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1850 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Elevated Pediatric Early Warning Score (PEWS) | 1 year
  frequency of patients whose PEWS score indicates 'risk for clinical deterioration' and receive a clinical intervention. PEWS 3 or greater (Scale is PEWS 0-6) is defined as at risk for clinical deterioration with a higher score concerning for worse clinical outcome.

SECONDARY OUTCOMES:
Time to antibiotics | 1 year
  Time to antibiotics defined as time from documented vital signs/PEWS to time of antibiotic administration measured in minutes
Time to IV fluid bolus | 1 year
  Time to fluids defined as time from documented vital signs/PEWS to time of documented IV fluid bolus measured in minutes
Volume of IV fluids | 1 year
  Volume of fluids received defined as volume given up to 60 minutes after the initiation of the first fluid bolus measured in milliliters
Length of stay | 1 year
  Length of stay for all patients admitted to the inpatient ward

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Niescierenko, MD MPH, Principal Investigator — Boston Children's Hospital
Locations (2):
- Palestinian Territories (2):
  - Beit Jala Hospital, Bethlehem
  - Rantisi Hospital, Gaza

IPD SHARING:
Plan to Share IPD: No